CLINICAL TRIAL: NCT02536586
Title: A Phase 1 Study of LY3023414 in Japanese Patients With Advanced Malignancies
Brief Title: A Study of LY3023414 in Japanese Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15838; I6A-JE-CBBH (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — LY3023414

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY3023414 (Experimental): LY3023414 administered orally, twice daily in 21-day cycles. Treatment will continue until disease progression, development of unacceptable toxicity, or other discontinuation criteria are met.
  Interventions: Drug: LY3023414

INTERVENTIONS:
Drug: LY3023414 — LY3023414 administered orally.

SUMMARY:
The main purpose of this study is to evaluate the tolerability of an investigational drug known as LY3023414 in Japanese participants with advanced cancer or cancer that has spread to another part(s) of the body. The study will also explore the safety of the drug. It will measure how much of the drug gets into the blood steam and how long the body takes to get rid of it. It will investigate anti-cancer activity.

ELIGIBILITY:
Inclusion Criteria

* Have histological or cytological evidence of a diagnosis of solid tumor that is advanced and/or metastatic and must be, in the judgment of the investigator, an appropriate candidate for experimental therapy after available standard therapies have failed or for whom standard therapy would not be appropriate.
* Have the presence of measurable or non-measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Have adequate organ and coagulation function.
* Have discontinued all previous cancer therapies, and any agents that have not received regulatory approval for any indication, for at least 21 days or 5 half-lives prior to study treatment, whichever is shorter, and recovered from the acute effects of therapy. Participants must have discontinued mitomycin-C or nitrosourea therapy for at least 42 days.
* Are able to swallow capsules.
* Males must agree to use medically approved barrier contraceptive precautions during the study and for 3 months following the last dose of study drug.
* Females with childbearing potential: Must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug, must have had a negative serum or urine pregnancy test ≤7 days before the first dose of study drug.
* A breastfeeding woman must not be breastfeeding. If a female who stops breastfeeding enters the study, breastfeeding must cease from the day of the first study drug administration until at least 3 months after the last administration.

Exclusion Criteria

* Have serious pre-existing medical conditions.
* Have symptomatic central nervous system malignancy or metastasis.
* Have known acute or chronic leukemia or current hematologic malignancies that, in the judgment of the investigator and sponsor, may affect the interpretation of results.
* Have a known active fungal, bacterial, and/or known viral infection.
* Intolerance to any previous treatment with any phosphatidylinositol 3-kinase (PI3K)/AKT/mammalian target of rapamycin (mTOR) inhibitor. Treatment with any PI3K/AKT/mTOR inhibitor must have discontinued for at least 21 days or 5 half-lives prior to first study drug administration, whichever is shorter, and participants must have recovered from the acute effects of therapy.
* Have a second primary malignancy that, in the judgment of the investigator, and sponsor may affect the interpretation of results.
* Participants with active alcohol abuse, as determined by the investigator.
* Have a history of heart failure according to New York Heart Association Class ≥3.
* Have corrected QT (QTc) interval of >470 milliseconds (msec) on screening electrocardiogram (ECG).
* Have insulin-dependent diabetes mellitus or a history of gestational diabetes mellitus.
* Have any evidence of clinically active interstitial lung disease (ILD).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with LY3023414 Dose-Limiting Toxicities (DLT) | Cycle 1 (21 days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Plasma Concentration-Time Curve (AUC) of LY3023414 | Predose Cycle 1 through predose Cycle 3. (Cycle = 21 days.)
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3023414 | Predose Cycle 1 through predose Cycle 3. (Cycle = 21 days.)
Proportion of Participants With Best Overall Response (OR) of Partial Response (PR) or Complete Response (CR) (Overall Response Rate [ORR]) | Baseline through study completion (estimated as up to five months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Tokyo